CLINICAL TRIAL: NCT03224949
Title: Comparison of ALD, NASH, and Healthy Control Patients
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Other Study IDs: 17-718
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: ALD - Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy controls
  Interventions: Other: Blood draw
- Alcoholic hepatitis
  Interventions: Other: Blood draw
- Alcoholic steatosis
  Interventions: Other: Blood draw
- Alcoholic cirrhosis without HCC
  Interventions: Other: Blood draw
- Nonalcoholic steatohepatitis (NASH)
  Interventions: Other: Blood draw
- Alcoholic cirrhosis with HCC
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Patients will have a one time blood draw

SUMMARY:
The availability of biological samples from individuals with alcoholic liver disease (ALD), as well as samples from appropriate heavy drinking, yet healthy controls and non-drinking healthy controls, is an essential first step in the translation of basic research advances to the clinic. The purpose of the Clinical Core component of the P50 Northern Ohio Alcohol Center (NOAC) is to provide biological samples (plasma/serum, buffy coats, and urine) from patients with different stages of alcoholic liver disease, as well as healthy control subjects, to members of the NOAC. These samples can then be used to test specific hypotheses related to the presence of specific biomarkers in the serum, functional immune activity in PBMCs and/or genetic polymorphisms that may predict severity of disease, short- and long-term morbidity and mortality and/or responsivity to specific therapeutic interventions commonly used in clinical practice. This study is building on the established biorepositories and the diversity of outstanding clinical expertise at the Cleveland Clinic. This biorepository included clinical samples (plasma, serum, buffy coats, and urine) from patients with different stages of ALD and subjects who are heavy drinkers without ALD, recruited from the Cleveland Clinic alcohol use disorder treatment clinic. This study will be responsible for collecting more data to help build the CCF-ALD biorepository via subject recruitment and communication and specimen collection.

ELIGIBILITY:
Alcoholic Steatosis Patients

Inclusion

* Fat accumulation (Steatosis) without signs of fibrosis/ inflammation in patients with alcohol abuse (alcohol intake >60 g/day in men and >40 g/day in women)
* Abnormal liver serum tests indicative of liver disease (elevated AST>ALT, y-glutamyl transpeptidase and bilirubin) .

Alcoholic Hepatitis with Mild Fibrosis

Inclusion

* Steatosis plus hepatocellular damage (presence of Mallory bodies and hepatocellular ballooning)
* Polymorphonuclear infiltrate
* Fibrosis stage 1-2

Alcoholic Hepatitis with Advanced Fibrosis

Inclusion

* Steatosis plus hepatocellular damage (presence of Mallory bodies and hepatocellular ballooning)
* Polymorphonuclear infiltrate
* Fibrosis stage 3-4.

Alcoholic Cirrhosis

Inclusion

* Fibrosis stage 4
* Presence of complications of cirrhosis such as esophageal varices with our without a previous episode of bleeding, splenomegaly, ascites, hepatic corroborate the diagnosis of cirrhosis.

Alcoholic Cirrhosis with HCC

Inclusion

-Diagnostic criteria of cirrhosis and established HCC. The diagnosis of HCC will be established based on histological confirmation or contrast-enhanced radiographic imaging according to the AASLD recommendations.

Exclusion

* BMI>35
* HBV
* Hemochromatosis
* Wilson's disease
* Autoimmune hepatitis
* Drug-inducted liver disease
* Hepatitis C
* Antitrypsin deficiency
* Patients who do not sign informed consent.

Non-alcoholic steatohepatitis

Inclusion -Biopsy proven NASH and chronic liver disease due to HCV patients.

Exclusion

* Cancer
* Diabetes
* Hypertension
* CAD or stroke
* Past history of liver disease
* Hepatitis C
* Antitrypsin deficiency
* Alcohol consumption of less than 7 drinks per week for women and less than 14 drinks per week for men
* BMI >35.

Healthy controls

Inclusion

-AUDIT-C score less than 4 in men and less than 3 in women.

Exclusion

* Cancer (except of non-melanoma skin cancer)
* Diabetes
* Hypertension
* Hypercholesterolemia
* Coronary artery disease or stroke
* History of current or past liver disease of any etiology
* BMI >27Kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from within Cleveland Clinic
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Biorepository | This is a 5 year study
  The goal of this study is to create a biorepository of samples from patients with different types of liver disease compared to each other and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Srinivisan Dasarathy, MD, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Helsley RN, Miyata T, Kadam A, Varadharajan V, Sangwan N, Huang EC, Banerjee R, Brown AL, Fung KK, Massey WJ, Neumann C, Orabi D, Osborn LJ, Schugar RC, McMullen MR, Bellar A, Poulsen KL, Kim A, Pathak V, Mrdjen M, Anderson JT, Willard B, McClain CJ, Mitchell M, McCullough AJ, Radaeva S, Barton B, Szabo G, Dasarathy S, Garcia-Garcia JC, Rotroff DM, Allende DS, Wang Z, Hazen SL, Nagy LE, Brown JM. Gut microbial trimethylamine is elevated in alcohol-associated hepatitis and contributes to ethanol-induced liver injury in mice. Elife. 2022 Jan 27;11:e76554. doi: 10.7554/eLife.76554. PMID 35084335